CLINICAL TRIAL: NCT05563961
Title: A Partial Randomized, Single-blind or Open-label, Dose-escalation With Multiple-dose Design Study to Evaluate the Pharmacokinetics of Acetaminophen and Its Toxic Metabolites With Panadol® and SafeTynadol® in Healthy Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinew Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: Oral AAP-002
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis; Pharmacology
Keywords: acetaminophen; acute liver failure
MeSH Terms: conditions — Hepatitis; Liver Failure, Acute | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Panadol (Active Comparator): • Cohort 1- 6 Subjects to receive oral Panadol® 4,000 mg (2 tablets Q6H, 4 dosages, 8 tablets or 4,000 mg)
  Interventions: Drug: Panadol®
- SafeTynadol® (Experimental): * Cohort 2- 6 Subjects to receive oral SafeTynadol® 4,000 mg (2 tablets Q6H, 4 dosages, 8 tablets or 4,000 mg)
  * Cohort 3- 6 Subjects to receive oral SafeTynadol® 4,500 mg (3 tablets at first dosage and 2 tablets at second to forth dosage Q6H, 4 dosages, 9 tablets or 4,500 mg)
  * Cohort 4- 6 Subjects to receive oral SafeTynadol® 5,000 mg (3 tablets at first to second dosage and 2 tablets at third to forth dosage Q6H, 4 dosages, 10 tablets or 5,000 mg)
  * Cohort 5- 6 Subjects to receive oral SafeTynadol® 6,000 mg (3 tablets Q6H, 4 dosages, 12 tablets or 6,000 mg)
  * Cohort 6- 6 Subjects to receive oral SafeTynadol® 8,000 mg (4 tablets Q6H, 4 dosages, 16 tablets or 8,000 mg)
  * Cohort 7- 6 Subjects to receive oral SafeTynadol® 10,000 mg (5 tablets Q6H, 4 dosages, 20 tablets or 10,000 mg)
  * Cohort 8- 6 Subjects to receive oral SafeTynadol® 12,000 mg (6 tablets Q6H, 4 dosages, 24 tablets or 12,000 mg)
  Interventions: Drug: SafeTynadol®

INTERVENTIONS:
Drug: Panadol® — Reference Drug. Multiple-dose stage: Cohort 1, 2 tablets Q6H (total 4 dosages, 8 tablets or 4,000 mg)
  Arms: Panadol
Drug: SafeTynadol® — Test Drugs. Multiple-dose stage:
  Cohort 2, 2 tablets Q6H (total 4 dosages, 8 tablets or 4,000 mg) Cohort 3, 3 tablets at first dosage and 2 tablets at second to forth dosage Q6H (total 4 dosages, 9 tablets or 4,500 mg) Cohort 4, 3 tablets at first to second dosage and 2 tablets at third to forth dosage Q6H (total 4 dosages, 10 tablets or 5,000 mg) Cohort 5, 3 tablets Q6H (total 4 dosages, 12 tablets or 6,000 mg) Cohort 6, 4 tablets Q6H (total 4 dosages, 16 tablets or 8,000 mg) Cohort 7, 5 tablets Q6H (total 4 dosages, 20 tablets or 10,000 mg) Cohort 8, 6 tablets Q6H (total 4 dosages, 24 tablets or 12,000 mg)
  Arms: SafeTynadol®

SUMMARY:
To investigate and compare the possible response of Panadol® and SafeTynadol® formulations in healthy volunteers and the safety in SafeTynadol® dose-limiting hepatotoxicity.

DETAILED DESCRIPTION:
Subjects will be randomized to Cohort 1 and cohort 2 in the study without crossover, Cohort 3-8 will be a dose-escalation manner. An effort will be made to balance the number of males and females in each cohort.

The first treatment cohort 1 and 2 will enroll 12 study volunteers. The volunteers of cohort 1 will receive Panadol® oral dosage form is 500 mg*2 tablets = 1,000 mg/ person every 6 hours daily of the multiple-dose treatment (Q6H, total 4 dosages, 8 tablets, 4,000 mg) (n = 6) and cohort 2 will receive SafeTynadol® oral dosage form is 500 mg*2 tablets = 1,000 mg/ person every 6 hours daily of the multiple-dose treatment (Q6H, total 4 dosages, 8 tablets, 4,000 mg) (n = 6) in an single-blind, randomized manner.

About one to three weeks later, cohorts 3-8 will be studied in an order of increasing dose of SafeTynadol® starting from 4,500 mg increment to a maximum dose of 12,000 mg of SafeTynadol® if the previous cohort do not meet the significant criteria of hepatotoxicity.

Cohort 3-8 will initially enroll 3 study volunteers. Volunteers will receive SafeTynadol® oral dosage form is 500 mg*3 tablets at first dosage (1500 mg) and 500 mg every 6 hours *2 tablets at second to fourth dosage (1000 mg) person every 6 hours daily of the multiple-dose treatment (Q6H, total 4 dosages, 9 tablets, 4,500 mg) at cohort 3 or Volunteers will receive SafeTynadol® oral dosage form is 500 mg*3 tablets at first and second dosage (1500 mg) and 500 mg every 6 hours *2 tablets at third and fourth dosage (1000 mg) person every 6 hours daily of the multiple-dose treatment (Q6H, total 4 dosages, 10 tablets, 5,000 mg) at cohort 4 or Volunteers will receive SafeTynadol® oral dosage form is 500 mg*3 tablets = 1,500 mg/ person every 6 hours daily of the multiple-dose treatment (Q6H, total 4 dosages, 12 tablets, 6,000 mg) at cohort 5 or Volunteers will receive SafeTynadol® oral dosage form is 500 mg*4 tablets = 2,000 mg/ person every 6 hours daily of the multiple-dose treatment (Q6H, total 4 dosages, 16 tablets, 8,000 mg) at cohort 6 or Volunteers will receive multiple doses of SafeTynadol® oral dosage form 500 mg every 6 hours * 5 tablets = 2,500 mg/person every 6 hours daily of the multiple-dose treatment (Q6H, 4 doses, 20 tablets, 10,000 mg) at Cohort 7 or Volunteers will receive multiple doses of SafeTynadol® oral dosage form 500 mg every 6 hours * 6 tablets = 3,000 mg/person every 6 hours daily of the multiple-dose treatment (Q6H, 4 doses, 24 tablets, 12,000 mg) at Cohort 8.

In Cohort 3-8, liver function tests will be administered two hours after the third dose to confirm that the hepatotoxicity criteria are not met before the fourth dose can be administered and Cohort 6-8 will perform liver function tests two hours after the second dose administered to confirm that the hepatotoxicity criteria are not met before the third dose can be administered. After 3 study volunteers to confirm that did not meet significant hepatotoxicity occurs then another 3 study volunteers were included, study will in a dose-escalation manner.

Except at admission blood blank sampling to Clinical Research Center on day 1 at 10:00, sampling will be obtained at the following times last post dose: 0 (prior to the last dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours after administration (21 samples) to assess acetaminophen concentrations and its metabolites concentrations. In addition, Cohort 1-8 blood sample for liver function test (ALT, AST, total bilirubinl) and PT(INR) will be obtained on day 1 (10:00) after admission, two hours after the third dose on day 2 and 24, 48, 72, 96, 120 and 144 hours after the last dose, Cohort 6-8 will increase the assessment of liver function tests two hours after the second dose. Blood samples for blood chemistry, PT(INR), hematology (CBC) and OGSP will be collected on 168 hours for post-study evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy adult subjects between 20-50 years of age.
* Body weight within 80-120% of ideal body weight.

  * Male Ideal body weight = (height - 80) x 0.7
  * Female Ideal body weight = (height - 70) x 0.6
* Acceptable medical history and physical examination including:
* normal ECG results within six months prior to dosing.
* no particular clinical significance in general disease history within two months prior to dosing.
* Acceptable clinical laboratory determinations without significant deviation from normal values within two months prior to dosing, which includes AST (SGOT), ALT (SGPT), r-GT, alkaline phosphatase, total bilirubin, albumin, glucose, BUN, uric acid, creatinine, total cholesterol, triglyceride (TG), PT(INR) and OGSP.
* Acceptable hematology within two months prior to dosing, which includes hemoglobin, hematocrit, red blood cells, MCV, MCH, MCHC, white blood cells, differential white blood cells and platelets.
* Acceptable urinalysis within two months prior to dosing, which includes pH, blood, glucose and protein.
* Signed the written informed consent to participate in this study

Exclusion Criteria:

* History or presence of alcohol abuse, defined as consumption of more than 210 mL of alcohol per week (the equivalent of 14 glasses of 120-mL wine or 14 cans of 350-mL beer), or other substance abuse within the prior two years.
* A clinically significant disorder involving the allergy, cardiovascular, respiratory, renal, gastrointestinal/hepatic, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the clinical investigator).
* History of allergic response(s) to acetaminophen, mannitol, sucralose or related drugs.
* History of clinically significant allergies including drug allergies or allergic bronchial asthma.
* Evidence of chronic or acute infectious diseases.
* Any clinically significant illness or surgery during the two month prior to dosing (as determined by the clinical investigator).
* Taking any drug known to induce or inhibit hepatic drug metabolism within one month prior to the beginning of the study.
* Receiving any investigational drug within one month prior to dosing.
* Taking any prescription medication or any nonprescription medication within two weeks prior to dosing.
* Donating greater than 150 ml of blood within two months prior to dosing or donating plasma (e.g. plasmapheresis) within two weeks prior to dosing.
* Consumption of caffeine, xanthine-containing products (i.e. coffee, tea, caffeine-containing sodas, colas and chocolate, etc.) and/or alcohol within 48 hours prior to days on which dosing is scheduled and during the periods when blood samples are being collected.
* Any other medical reason as determined by the clinical investigator.
* Subject is pregnant or breastfeeding.
* Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, intrauterine device (IUD), barrier device or abstinence) throughout the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ALT level within study periods | Day 1-9

SECONDARY OUTCOMES:
Incidence of peak ALT elevations > 1X ULN within study periods | Day 1-9
Incidence of peak ALT elevations > 2X ULN within study periods | Day 1-9
Incidence of peak ALT elevations > 3X ULN within study periods | Day 1-9
Incidence of peak ALT elevations > 5X ULN within study periods | Day 1-9
Incidence of peak ALT elevations > 8X ULN within study periods | Day 1-9
Incidence of total bilirubin > 2.5mg/dL within study periods | Day 1-9
Incidence of PT (INR) > 1.25 within study periods | Day 1-9
Hepatic failure rate | Day 1-9
  Hepatic failure rate (hepatic encephalopathy, ascites, total bilirubin >2.5mg/dL, PT(INR) >1.25 , or liver transplantation) within study periods
Free plasma acetaminophen-cysteine (AAP-Cys) and AAP-Cys adducts | Day 1-9
  The time-interval weighted area under the curve (AUC) of free plasma acetaminophen-cysteine (AAP-Cys) and AAP-Cys adducts within study periods
The time-interval weighted area under the curve (AUC) of ALT level within study periods | Day 1-9

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided